CLINICAL TRIAL: NCT05913414
Title: A Randomised Phase II Trial of Iron Isomaltide Versus Oral Iron Supplement for Radiotherapy or Chemotherapy Associated Iron-deficiency Anemia Patients With Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Iron Isomaltide for Iron-deficiency Anemia Patients With Locally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-747-01
Record Dates: First submitted 2023-04-23; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma; Iron-deficiency; Anemia
Keywords: Nasopharyngeal Carcinoma; iron-deficiency anemia
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Anemia, Iron-Deficiency; Anemia | interventions — iron isomaltoside 1000; Niferex; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Iron Isomaltide (Experimental): Patients receive iron Isomaltide after anti-tumor therapy.
  Interventions: Drug: Iron Isomaltoside 1000; Radiation: Intensity-modulated radiotherapy
- Oral iron supplement (Active Comparator): Patients receive polysaccharide iron complex after anti-tumor therapy.
  Interventions: Drug: Polysaccharide Iron Complex Pill; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Iron Isomaltoside 1000 — Patients receive Iron isomaltoside after IC and CCRT
  Other Names: Iron isomaltoside
  Arms: Iron Isomaltide
Drug: Polysaccharide Iron Complex Pill — Patients receive Polysaccharide Iron Complex Pill after IC and CCRT
  Arms: Oral iron supplement
Radiation: Intensity-modulated radiotherapy — All patients received intensity-modulated radiotherapy before enrolled.

SUMMARY:
Primary purpose： To evaluate the difference of hematopoietic response rate at 1 month after concurrent chemoradiotherapy between iron isomaltide and oral iron supplement for treating iron-deficiency anemia patients with locally advanced nasopharyngeal carcinoma.

Secondary purpose:

To evaluate the difference of hematopoietic response rate, tolerance, acute side effects, qualtiy of life at 2 months and 3 months after concurrent chemoradiotherapy between Iron Isomaltide and oral iron supplement for treating iron-deficiency anemia patients with locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Iron-deficiency anemia patients with locally advanced nasopharyngeal carcinoma will be enrolled and receive iron Isomaltide or oral iron supplement after randomised. The hematopoietic response rate, tolerance, acute side effects, qualtiy of life and long time survival would be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer and sign the informed consent in person.
* Aged 18-65
* Pathological diagnosis of non-keratinizing NPC (differentiated or undifferentiated, as WHO II, III type).
* Clinical stage of III-IVA（8thAJCC/UICC staging system）
* Complete induction chemotherapy and concurrent chemoradiotherapy.
* With ECOG score 0-1.
* Female subjects: surgical sterilization or postmenopausal patients, or agree to use a medical approved contraceptive measure such as Intrauterine device (IUD), contraceptives or condoms during the study period.
* HGB <130g/L(male)，HGB<120g/L(female).
* Serum ferritin≤800ug/L。
* Liver function: ALT, AST < 2.5 times the upper limit of normal (ULN), total bilirubin < 2.0 × ULN;
* Renal function: serum creatinine <1.5×ULN.

Exclusion Criteria:

* Recurrence or distant metastasis nasopharyngeal carcinoma.
* Keratinizing squamous cell carcinoma (WHO type I).
* Pregnant or breastfeeding women, who are in their childbearing years and have not used effective contraception.
* Previous or concurrently with other malignancies, exclude cured skin basal cell carcinoma and cervical carcinoma in situ.
* Patients with severely diminished functions of the heart, liver, lung, kidney and bone marrow;
* Serious, unmanaged medical conditions and infections.
* Those with other therapeutic contraindications.
* Use of other investigational medications or clinical studies concurrently.
* Refused or incapacity to sign the informed consent to participate in the study.
* People having mental or personality disorders, disability, or limited civil capacity.
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.
* HGB>130g/L(male)，HGB >120g/L(female).
* Received transfusion therapy before.
* Receipt of oral or IV iron supplements or ESAs up to 4 weeks before inclusion
* Ferritin > 800 ng/ml
* Ongoing bleeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Hematopoietic response rate | 1 month
  Hematopoietic response rate at one month after IC+CCRT.

SECONDARY OUTCOMES:
Hematopoietic response rate | 2 month
  Hematopoietic response rate at two months after IC+CCRT.
Hematopoietic response rate | 3 month
  Hematopoietic response rate at three months after IC+CCRT.
Acute side effects | 1 month
  The acute side effects of iron isomaltide
Quality of life scores | 1 month
  The scores of each scale of quality of life questionaires for FACT-An
The difference of HGB | 1,2,3 months
  The difference of HGB after patients receiving iron supplements
The score of concise fatigue scale | 1,2,3 months
  Calculated by Concise fatigue scale
The difference of serum iron | 1,2,3 months
  The difference of HGB after patients receiving iron supplements

CONTACTS AND LOCATIONS:
Overall Officials: Shan Shan Guo, Dr, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No